CLINICAL TRIAL: NCT02389231
Title: " Anemil Trial ": Phase I/II Clinical Trial Evaluating the Interest of Interleukine-2 for Patients With Active Warm Hemolytic Anemia Resistant to Conventional Treatment
Brief Title: Evaluating the Interest of Interleukine-2 for Patients With Active Warm Hemolytic Anemia Resistant to Conventional Treatment
Acronym: ANEMIL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2013/29
Record Dates: First submitted 2015-02-13; First posted 2015-03-17 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Autoimmune Hemolytic Anemia
Keywords: interleukine 2; warm autoimmune hemolytic anemia; CD8 regulatory T cells
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low doses of Interleukine-2 (Experimental): Low doses of Interleukine-2 over a 9 week treatment period
  Interventions: Drug: Interleukine-2

INTERVENTIONS:
Drug: Interleukine-2 — Four courses of IL2 ( [Proleukin, Novartis]) will be administered subcutaneously for 5 days.
  The first course will be limited to a dose of 1.5 million IU per day and followed by a 9 day wash-out.
  The other courses of 3 million IU per day will be initiated after a 16 day wash-out.
  Other Names: PROLEUKIN 18M; aldesleukine

SUMMARY:
The investigators have demonstrated that the mean percentage of circulating CD8+ regulatory T (CD8 Tregs) cells is significantly higher in patients with warm hemolytic anemia (wAHAI) in remission than in controls and is correlated to hemoglobin levels. In vitro, low dose of interleukine-2 (IL2) induce the expansion of CD8 Tregs. The objective is to demonstrate that, over a 9 week treatment period; low doses of IL2 can induce the expansion of CD8Tregs in patients with active wAHAI.

DETAILED DESCRIPTION:
wAIHA is a B-cell-mediated autoimmune disease in which red blood cells are targeted by autoantibodies, which leads to marked decrease in their lifespan. The investigators demonstrated two years ago in a multivariate retrospective study that the CD3+CD8+ HLA-DR+ T-cell population was associated to a better outcome. The investigators observed that the proportion of circulating CD3+CD8+CD25highFoxp3+ T cells was significantly higher in patients with wAIHA in remission than in controls and correlated to hemoglobin levels. Extensive phenotyping and functional analysis revealed that those cells were bona fide Tregs acting in an IL10-dependent manner. Finally, culture of PBMC from normal donors or active wAIHAI patients with low dose of IL2 promoted the expansion of functional CD3+CD8+CD25+Foxp3+. Those observations constituted the rationale to propose low dose of IL2 to treat patients with active wAIHA with the objective of demonstrating that this treatment is able to induce the expansion of CD8Tregs, over a 9 week treatment period.

Four courses of IL2 (aldesleukin [Proleukin, Novartis]) will be administered subcutaneously for 5 days. The first course will be limited to a dose of 1.5 million IU per day and followed by a 9 day wash-out. The other courses of 3 million IU per day will be initiated after a 16 day wash-out.

Patients will be evaluated on day 1 and day 5 of each treatment course, before the first and last administration of interleukin-2 and will also be evaluated at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old)
* wAHAI defined by the presence of hemolysis and positive coombs test (IgG +/-C3)
* Absence of infection or other hematologic disease
* wAHAI not responding to conventional steroids despite a dose over 10 mg
* No treatment with rituximab for a minimum of 6 months
* Signed informed consent form

Exclusion Criteria:

* Less than 18 years old
* Cold AHAI
* IL2 allergy
* Chemiotherapy or immunosuppressive treatment
* Treatment with rituximab for less than 6 months
* Neoplasia or hematologic malignancy
* Aplastic anemia
* Neutropenia ≤ 1000 mm3
* Infection
* Hepatitis B or C
* wAHAI associated with systemic lupus erythematosus depending on ACR criteria
* Cardiac insufficiency
* Hypertension
* Pulmonary insufficiency
* Liver cirrhosis
* Thrombopenia below 50000/mm3
* Drug addiction, alcohol abuse
* Psychiatric disorder
* Absence of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Percentage of LTCD8+CD25highFoxp3+ . | 9 weeks after inclusion
  Increase of the percentage of LTCD8+CD25highFoxp3+ at the end of the IL2 treatment.

SECONDARY OUTCOMES:
Incidence of complications with the treatment. | 6 months after inclusion
  Safety of the treatment during the trial and 6 months after the inclusion
Hemolysis as measured by hemoglobin, haptoglobin, reticulocytes and LDH levels | 5 days, 20 days, 40 days, 61 days, 63 days and 6 months after inclusion
  Impact of IL2 on hemolysis defined by hemoglobin, haptoglobin, reticulocytes, LDH levels
Evaluation of lymphocyte sub-populations | 5 days, 20 days, 40 days, 61 days, 63 days and 6 months after inclusion
  Impact of IL2 on lymphocyte sub-populations (NK cells, B lymphocyte, CD4T lymphocyte, CD8T lymphocytes, CD4Tregs levels) at each time point of evaluation.
Evaluation of lymphocyte activation. | 5 days, 20 days, 40 days, 61 days, 63 days and 6 months after inclusion
  Impact of IL2 on lymphocyte activation defined by DR expression at each time point of evaluation.
Dose of steroid treatment | 5 days, 20 days, 40 days, 61 days, 63 days and 6 months after inclusion
  Impact of IL2 on steroid treatment (dose) during the trial and 6 months after the inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Estibaliz LAZARO, Prof, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, Prof, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux Hôpital Haut Lévêque, Pessac, Aquitaine, France